CLINICAL TRIAL: NCT03752554
Title: Assessment of Neurosensory Function Following Segmental Mandibular Resection of Non-malignant Lesions With Inferior Alveolar Nerve Preservation: A Case Series Trial
Brief Title: Assessment of Neurosensory Function Following Segmental Mandibular Resection.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, sherif awad, assistant researcher in national research centre, Cairo University
Other Study IDs: CEBD-CU-2018-11-10
Record Dates: First submitted 2018-11-17; First posted 2018-11-26 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2018-12

CONDITIONS: Resection Cavity
Keywords: segmental mandibular resection-IAN
MeSH Terms: interventions — Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: segmental resection — All cases will undergo surgery under general anesthesia. The mandibular lesion will be segmentally resected. The cuts will be performed with the aid of the prefabricated digital template. The neurovascular bundle will be separated and protected. Then reconstruction will be performed

SUMMARY:
This study wInclusion criteria for this study will be as follows:

* Age group: from 15 to 60 years old.
* Patients with with non malignant mandibular neoplasms indicated for segmental resection.

Exclusion criteria:

* Patients with malignant mandibular neoplasms.

All cases will undergo surgery under general anesthesia. The mandibular lesion will be segmentally resected. The cuts will be performed with the aid of the prefabricated digital template. The neurovascular bundle will be separated and protected. Then reconstruction will be performed.

Postoperative patient evaluation:

Neurosensory examination:

Assessment of the inferior alveolar nerve function will be performed preoperatively, 2 and 12 weeks postoperatively through Trigeminal somatosensory evoked potential technique. Six months postoperatively by CBCT for assessment of recurrence

DETAILED DESCRIPTION:
This study will include 10 patients complaining from non malignant mandibular lesions. nopatients will be selected from the outpatient clinic of the Oral & Maxillofacial Surgery department, faculty of Dental Medicine Cairo University.

All the procedures will be explained for all patients before undergoing operation and informed consent process will be taken, this study will be displayed to the research ethics committee to obtain approval.

Inclusion criteria for this study will be as follows:

* Age group: from 15 to 60 years old.
* Patients with with non malignant mandibular neoplasms indicated for segmental resection.

Exclusion criteria:

* Patients with malignant mandibular neoplasms. 1- Pre-operative phase

Patients will be subjected to:

Case history including personal data, medical, a-surgical and family history b-Clinical examination c.Radiographic examination using orthopantogram, and computed tomography (CT) Preoperative anesthesia assessment for fitness for general anesthesia.d Treatment planning and fabrication of the digital template.e 2 -Operative phase All cases will undergo surgery under general anesthesia. The mandibular lesion will be segmentally resected. The cuts will be performed with the aid of the prefabricated digital template. The neurovascular bundle will be separated and protected. Then reconstruction will be performed.

3-Postoperative care:

Postsurgical instructions and follow up:

Proper postoperative instructions will be given the patient, in addition to the postoperative medications including antibiotics, corticosteroids and analgesics.

Postoperative patient evaluation:

Neurosensory examination:

Assessment of the inferior alveolar nerve function will be performed preoperatively, 2 and 12 weeks postoperatively through Trigeminal somatosensory evoked potential technique. Six months postoperatively by CBCT for assessment of recurrence.

Statistical analysis:

Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 21 (SPSS Inc. Chicago). The data will be compared using paired t-test.

ELIGIBILITY:
Inclusion Criteria:

* -Age group: from 15 to 60 years old.
* Patients with with non malignant mandibular neoplasms indicated for segmental resection..

Exclusion Criteria:

* -Patients with malignant mandibular neoplasms

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients with non malignant mandibular lesions
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
measurement of nerve stimulation | 3 months
  somatosensory evoked potential technique

CONTACTS AND LOCATIONS:
Overall Officials: ragia mo mounir, professor, Principal Investigator — kaser elany cairo univeristy
Locations (1):
- Kasr Al Einy Cairo Univeristy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
international publishing

REFERENCES:
- See also: preservation of inferior alveolar nerve — https://www.ncbi.nlm.nih.gov/pubmed/?term=Preservation+of+the+inferior+alveolar+neurovascular+bundle+in+the+osteotomy+of+benign+lesions+of+the+mandible+using+a+digital+template.